CLINICAL TRIAL: NCT07004296
Title: A Phase Ia/Ib Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Antitumor Activity of HDM2005 in Patients With Advanced Solid Tumors
Brief Title: A Study of HDM2005 in Patients With Advanced Solid Tumor
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hangzhou Zhongmei Huadong Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HDM2005-103
Record Dates: First submitted 2025-05-27; First posted 2025-06-04 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-05

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- HDM2005 (Experimental): In dose escalation phase, participants will be administered escalating doses of HDM2005 at 1.8~2.5mg/kg IV on Day 1 of repeated 21-day cycles or 1.2~2.0mg/kg IV on Day 1 of repeated 14-day cycles .
  In dose expansion phase, participants will be administered to recommended dose for expansion (RDE) of HDM2005 .
  Interventions: Drug: HDM2005

INTERVENTIONS:
Drug: HDM2005 — HDM2005 will be administered via IV infusion.

SUMMARY:
This is a study evaluating the efficacy, safety, and pharmacokinetics ofHDM2005 in participants with metastatic solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Agree to follow the study treatment protocol and visit schedule, enroll voluntarily and sign a written informed consent.
2. Male or female aged ≥ 18 years at the time of signing the ICF;
3. ECOG performance status of 0-1.
4. Life expectancy of at least 3 months.
5. Specific types of advanced solid tumors that have been confirmed by histopathological examination.
6. Has metastatic disease that has progressed during or following previous treatment appropriate for the disease type.
7. All subjects are required to provide archived tissue (5 unstained sections) obtained within the previous 2 years or fresh tissue for ROR1 expression testing at the central laboratory.
8. Presence of radiographically measurable disease.
9. Subjects must have recovered (to ≤ Grade 1) from any AE associated with prior anticancer therapy.
10. Has adequate organ function.
11. Female subjects of childbearing potential should agree to use contraception methods during the study and for 6 months after the end of the study; have a negative serum pregnancy test within 7 days before study enrollment; and male subjects should agree to use contraceptive avoidance measures during the study and for 6 months after the end of the study.

Exclusion Criteria:

1. Patients with active brain metastases (defined as stable for < 4 weeks, or symptomatic, or requiring antiepileptic drug/hormonal therapy, or meningeal metastases).
2. Subjects have another primary malignancy ,with the following exceptions: adequately treated non-melanoma skin cancer without evidence of disease recurrence and adequately treated carcinoma in situ without evidence of disease recurrence,et al.
3. History of severe bleeding disorders .
4. History of chronic pancreatitis or acute pancreatitis within 6 months.
5. History of interstitial lung disease, radiation pneumonitis requiring steroid therapy, or any evidence of clinically active interstitial lung disease.
6. Patients with uncontrolled pleural effusion, pericardial effusion or ascites requiring repeated drainage after intubation and drainage,VEGF inhibitors, platinum and other drugs injection (subjects with stable symptoms for at least one week after treatment can be enrolled).
7. Prior solid organ transplantation.
8. Has peripheral neuropathy of Grade >1.
9. Has significant cardiovascular or cerebrovascular diseases.
10. Has an uncontrolled ongoing infection.
11. Active infectious disease, such as HIV infection, active hepatitis B, active hepatitis C (positive RNA result), active syphilis.
12. Receiving corticosteroids (prednisone equivalent more than10 mg/day).
13. Contraindication to any component of HDM2005.
14. History of drug anaphylactic shock, severe food allergy, uncontrolled asthma or COPD.
15. Female subjects who are pregnant, lactating or planning to become pregnant during the study.
16. Known history of mental illness or substance abuse that would impair the subject's ability to cooperate with study requirements.
17. Prior or current evidence of any disease, treatment, or laboratory abnormality that, in the opinion of the investigator, could affect the outcome of the study, prevent the subject from participating in the study entirely, or is not in the subjects' best interest.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-05-29 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicity (DLT) events (for dose escalation phase) | up to 21 days or 28 days following first dose
  DLT will be determined by definition during the DLT observation period.
Incident and severity of adverse events(for dose escalation phase) | Until 28 days after the last dose or initiation of a new antineoplastic therapy, whichever occurs first.
  The safety profile of HDM2005 will be assessed by monitoring the adverse events (AE) per the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0.
Progression-free survival(PFS)(for dose expansion phase) | Approximately 30 months
  PFS, defined as the interval from the start of study treatment to the earlier of the first documentation of disease progression or death from any cause per RECIST, Version 1.1.
Objective Response Rate (ORR)(for dose expansion phase) | Approximately 18 months
  Objective response rate (ORR), which includes best response of complete response (CR) or partial response (PR) as assessed by the investigator.
Recommended Phase 2 Dose (RP2D) (for dose expansion phase) Recommended Phase 2 Dose (RP2D) (for dose expansion phase) Recommended Phase 2 Dose (RP2D) (for dose expansion phase) | Approximately 30 months
  The selection of RP2D will be based on consideration of overall safety information together with available pharmacokinetic,E-R relationships, and efficacy data. The selection of RP2D will be based on consideration of overall safety information together with available pharmacokinetic and efficacy data.

SECONDARY OUTCOMES:
Plasma concentration of HDM2005, total antibody and the free MMAE | up to 28 days following last dose
  Plasma concentration of HDM2005, total antibody and the free MMAE will be reported for each arm.
Immunogenicity | up to 28 days following last dose
  Number and percentage of anti-drug antibody (ADA)-positive patients will be assessed.
Objective Response Rate (ORR)(for dose escalation phase) | Approximately 18 months
  Objective response rate (ORR), which includes best response of complete response (CR) or partial response (PR) as assessed by the investigator.
Time to Response (TTR) | Approximately 30 months
  TTR is defined as the interval from the start of study therapy to the first documentation of an objective response.
Duration of Response (DOR) | Approximately 30 months
  DOR is defined as the interval from the first documentation of objective response to the earlier of the first documentation of disease progression/relapse or death from any cause.
Overall survival (OS) | Approximately 30 months
  OS is defined as the interval from the start of study therapy to death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University shanghai Cancer Center, Shanghai, Shanghai Municipality, China